CLINICAL TRIAL: NCT05709197
Title: The Effectiveness of Adding Braun Anastomosis to Standard Child Reconstruction to Reduce Delayed Gastric Emptying After Pancreatoduodenectomy (REMBRANDT): a Multicenter Randomized-controlled Trial
Brief Title: The Effectiveness of Adding Braun Anastomosis to Standard Child Reconstruction After Pancreatoduodenectomy
Acronym: REMBRANDT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL 82918.091.22
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Disease; Pancreatic Cancer; Delayed Gastric Emptying
Keywords: Randomized controlled trial; Prospective studies; Braun anastomosis; Braun enteroenterostomy
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Neoplasms; Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded considering their treatment allocation. The house officer, ward nurses and data managers who extract data concerning the primary and secondary endpoint will be blinded for the allocation as well. For this reason, this will be a patient- and observer blinded RCT.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Braun anastomosis (Experimental): Open pancreatoduodenectomy with Braun enteroenterostomy
  Interventions: Procedure: Braun anastomosis
- Standard Child reconstruction (Other): Open pancreatoduodenectomy only
  Interventions: Procedure: Standard Child reconstruction

INTERVENTIONS:
Procedure: Braun anastomosis — Participants will undergo open pancreatoduodenectomy (PD). The reconstruction technique will not be standardized. In addition to the reconstruction technique used, a side-to-side anastomosis will be created between the afferent and efferent jejunal limbs of the gastrojejunostomy (GJ) at 20 cm distance from the GJ. The anastomosis will be hand-sewn with monofilament PDS 3-0 one-layer running suture.
  Arms: Braun anastomosis
Procedure: Standard Child reconstruction — Participants will undergo open pancreatoduodenectomy (PD). The reconstruction technique will not be standardized. The surgeon is able to perform the PD as normally would be done (antecolic, retrocolic, pylorus-preserving or with distal gastric resecting).
  Arms: Standard Child reconstruction

SUMMARY:
The goal of this clinical trial (REMBRANDT) is to evaluate the effectiveness of adding an extra connection (i.e. 'Braun anastomosis') after standard reconstruction in pancreatic head resection in reducing the incidence of delayed gastric emptying.

DETAILED DESCRIPTION:
Rationale/hypothesis: The addition of Braun enteroenterostomy (BE) reduces the incidence of delayed gastric emptying (DGE) resulting in lower morbidity and healthcare costs after pancreatoduodenectomy.

Objective: To assess the effectiveness of adding BE in reducing DGE in patients undergoing open pancreatoduodenectomy.

Study design: A multicenter, patient and observer blinded, registry-based randomized controlled trial.

Study population: Patients undergoing an open pancreatoduodenectomy for all indications.

Intervention: Braun enteroenterostomy (BE), or Braun anastomosis, in addition to usual care.

Usual care/comparison: Pancreatoduodenectomy with standard Child reconstruction.

Main endpoints:

1. Incidence of DGE Grade B/C (according to International Study Group of Pancreatic Surgery (ISGPS)
2. Incidence of postoperative pancreatic fistulas (POPF) Grade B/C (according to ISGPS), anastomotic leak, complications, hospital length of stay, functional outcome at 12 months, in-hospital mortality, 30-day mortality, healthcare costs.

Sample size: 256 in total, 128 per arm

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients undergoing open pancreatoduodenectomy have an increased risk of postoperative complications such as DGE, POPF and anastomotic leak. The addition of BE, which is an anastomosis, could also result in a leak. However, this risk is diminishable compared to the risks of DGE and DGE related other complications like anastomotic leaks associated with standard pancreatoduodenectomy. Moreover, previous cohort studies involving BE do not describe an increased risk of adverse outcomes for BE.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing open pancreatoduodenectomy
* Provided informed consent
* Age over 18 years

Exclusion Criteria:

* Insufficient control of the Dutch language to read the patient information and to fill out the questionnaires in Dutch hospitals
* Previous bariatric surgery (such as Roux-en-Y gastric bypass, gastric sleeve)
* Pregnancy
* Bowel motility disorders
* Minimally invasive pancreatoduodenectomy
* Gastric outlet syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Delayed gastric emptying (DGE) | During hospitalization
  DGE is defined by the need for maintenance of the nasogastric tube (NGT), need for reinsertion of NGT for persistent vomiting after postoperative day (POD) 7, or inability to tolerate a solid diet.

SECONDARY OUTCOMES:
Pancreatic fistula (POPF) | During hospitalization
  Any measurable volume of drain output with an amylase level of more than 3 times the upper limit of normal serum amylase and clinically relevant condition or development of the patient directly related to the POPF.
Anastomotic leak | During hospitalization
  Anastomotic leaks of the hepatojejunostomy (HJ) or Braun enteroenterostomy (BE).
  Anastomotic leaks of the HJ manifest as bile leakage. This is defined as "fluid with an increased bilirubin concentration in the abdominal drain or in the intra-abdominal fluid on or after postoperative day 3, or as the need for radiologic intervention because of biliary collections or relaparotomy resulting from bile peritonitis. Increased bilirubin in the drain is defined as bilirubin concentration more than 3 times greater than the serum bilirubin concentration.
  An anastomotic leak of the BE is present when an abdominal CT with contrast shows leakage of contrast from the BE or when during relaparotomy dehiscence of the BE is apparent.
Postoperative complications: incidence and severity | During hospitalization
  Scored according to the modified Clavien-Dindo classification for surgical complications. Grade III and higher are considered clinically relevant in this study.
Number of days participants were hospitalized | During hospitalization
  The time period in days between hospital admission and discharge from the hospital.
Number of participants with in-hospital mortality | During hospitalization
  Any death during hospital admission.
30-day mortality | 30 days
  Any death occurring 30 days after pancreatoduodenectomy.
Quality of life (QoL) based on five dimensions | Change from baseline at 1 week, at 2 weeks, and 3 months
  The EQ-5D-5L standardized questionnaire will be used.
Participants perceived disease and treatment related quality of life | Change from baseline at 2 weeks, 3 months, and 12 months
  The European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30/PAN26 standardized quality of life questionnaires will be used.
Quality of recovery | Change from baseline at 1 week, at 2 weeks, and 3 months
  The QoR-15 standardized questionnaire will be used.
Functional outcome at 12 months | 12 months
  Participants will be phoned to assess whether they have complaints of delayed gastric emptying ("afferent loop syndrome").

CONTACTS AND LOCATIONS:
Overall Officials: Martijn WJ Stommel, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (12):
- Netherlands (12):
  - Amsterdam UMC, Amsterdam
  - OLVG, Amsterdam
  - Catharina hospital, Eindhoven
  - Medical spectrum Twente, Enschede
  - Groningen UMC, Groningen
  - Medical center Leeuwarden, Leeuwarden
  - LUMC, Leiden
  - Maastricht UMC+, Maastricht
  - St Antonius hospital, Nieuwegein
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - Isala hospital, Zwolle

REFERENCES:
- [Derived] Strijbos BTM, Hopstaken JS, Endo C, de Vries M, Atsma F, Adang E, van der Wees P, Besselink MGH, van Santvoort H, den Dulk M, Groot Koerkamp B, Mieog JSD, Zeverijn S, van Laarhoven CJHM, Stommel MWJ; Dutch Pancreatic Cancer Group. The effectiveness of adding Braun anastomosis to standard Child reconstruction to reduce delayed gastric emptying after pancreatoduodenectomy (REMBRANDT): study protocol for a multicentre randomised-controlled trial. Trials. 2025 Oct 2;26(1):387. doi: 10.1186/s13063-025-09051-x. PMID 41039614